CLINICAL TRIAL: NCT03259867
Title: Phase IIA Single-Arm Study of Treatment of Patients With Advanced Liver Cancer With a Combination of TATE (Transarterial Tirapazamine Embolization) Followed by an Anti-PD-1 Monoclonal Antibody
Brief Title: Combination of TATE and PD-1 Inhibitor in Liver Cancer
Acronym: TATE-PD1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teclison Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT-004
Record Dates: First submitted 2017-08-16; First posted 2017-08-24 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma; Gastric Cancer
Keywords: Hepatocellular carcinoma; Immune checkpoint inhibitor; Gastric cancer; Progression
MeSH Terms: conditions — Carcinoma, Hepatocellular; Stomach Neoplasms; Disease Progression | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: One arm for advanced HCC, and one for second line metastatic gastro-esophageal cancer . All enrolled patients will receive the same treatment with TATE and a PD-1 inhibitor (nivolumab) until disease progression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Advanced Hepatocellular carcinoma (Experimental): PD-1 inhibitor (Nivolumab 360 mg Q3W IV ) starts at day 1, and continues until progression.
  TATE treatment starts at day 8 for debulking up to 4 cycles. If escape lesion appears, two more TATE treatments can be given. Tirapazamine dose at 35 mg flat dose given before embolization.
  Interventions: Drug: Nivolumab Injectable Product; Combination Product: Trans-arterial tirapazamine embolization
- Metastatic Gastro-esophageal cancer (Experimental): PD-1 inhibitor (Nivolumab 360 mg Q3W IV) starts at day 1, and continues until progression.
  TATE treatment starts at day 8 for debulking up to 4 cycles. If escape lesion appears, two more TATE treatments can be given. Tirapazamine dose at 35 mg flat dose given before embolization.
  Interventions: Drug: Nivolumab Injectable Product; Combination Product: Trans-arterial tirapazamine embolization

INTERVENTIONS:
Drug: Nivolumab Injectable Product — a PD-1 immune check inhibitor
  Other Names: OPDIVO
Combination Product: Trans-arterial tirapazamine embolization — Embolization with Lipiodol and Gelfoam

SUMMARY:
This is a multi-center, open-label phase IIA study that investigates the preliminary efficacy of Trans-arterial Tirapazamine Embolization (TATE) treatment of liver cancer followed by a PD-1 checkpoint inhibitor (nivolumab). Patients with two types of cancers will be enrolled, advanced hepatocellular carcinoma (HCC),and metastatic gastric cancer. All enrolled patients need to have liver lesions and have progressed on a prior immune checkpoint inhibitor.

DETAILED DESCRIPTION:
The goal of the study is to investigate whether tumor necrosis induced by Trans-arterial Tirapazamine Embolization (TATE) treatment can boost anti-tumor immunity and enhance the therapeutic efficacy of immune checkpoint inhibitor. Patients with advanced liver cancers (primary HCC or metastatic gastric cancer) who have progressed on a prior immune checkpoint inhibitor will be enrolled in the study. Liver lesions will be treated with up to 4 TATE treatments for optimal debulking, which also serve as a vaccination process toward tumor. Lesion not treated with TATE will be used for monitoring the response toward a PD-1 inhibitor (Nivolumab) for abscopal effect. If a patient subsequently develops an "escape" to the PD-1 inhibitor, patient can have another 2 TATE treatments of the escaped tumor lesion. Dosing of the PD-1 inhibitor is per standard FDA-approved dosing schedule and continues until progressive disease. The efficacy will be assessed by the response rate (RR) using RECIST.

ELIGIBILITY:
1. Patients with a confirmed diagnosis of (1) advanced HCC or (2) metastatic gastric cancer.
2. Patients between ages 18 and 80
3. If HCC patients, they should have progressive disease (PD) on an immune therapy for advanced HCC. For patients with metastatic gastric cancer, they should have failed at least one line of systemic chemotherapy and an immune checkpoint inhibitor.
4. Patients with liver tumor lesions with at least one with a diameter of 2 cm or bigger, which is amendable for (super-)selective TATE as the target lesion.
5. ECOG score 2 or less
6. Child-Pugh scores 5-7 for HCC patients
7. All prior chemotherapy at least 4 weeks prior to study treatment. Immunotherapy not subject to this limitation.
8. No major GI bleeding in the prior 2 months.

8. Hgb>=8, platelet >= 50,000, Cr =< 2, AST and ALT < 10 X ULN, t-Bilirubin < 3, 9. Patients with a history of major autoimmune disorders excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | up to 24 months
  Per RECIST 1.1 criteria

SECONDARY OUTCOMES:
Duration of Response | up to 24 months
  From the date of image-demonstrated response to the date of progression
Time to Progression | up to 24 months
  From randomization to disease progression or death
Progression Free Survival | up to 24 months
  From randomization to disease progression or death
Overall survival | through study completion, an average of 3 years
  From randomization to death

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Abi-Jaoudeh, MD, Principal Investigator — UC Irvine Medical Center
Locations (3):
- United States (3):
  - University of California, Irvine, Orange, California
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu CH, Peng CM, Hwang JI, Liang PC, Chen PJ, Abi-Jaoudeh N, Giiang LH, Tyan YS. Phase I Dose-Escalation Study of Tirapazamine Chemoembolization for Unresectable Early- and Intermediate-Stage Hepatocellular Carcinoma. J Vasc Interv Radiol. 2022 Aug;33(8):926-933.e1. doi: 10.1016/j.jvir.2022.04.031. Epub 2022 Apr 30. PMID 35504436
- [Background] Abi-Jaoudeh N, Dayyani F, Chen PJ, Fernando D, Fidelman N, Javan H, Liang PC, Hwang JI, Imagawa DK. Phase I Trial on Arterial Embolization with Hypoxia Activated Tirapazamine for Unresectable Hepatocellular Carcinoma. J Hepatocell Carcinoma. 2021 May 17;8:421-434. doi: 10.2147/JHC.S304275. eCollection 2021. PMID 34041204